CLINICAL TRIAL: NCT00394069
Title: A Randomized, 3-Period, Multiple-Dose, Multicenter Study to Evaluate the Safety, Tolerability, and Plasma Concentration Profile of Montelukast Administered Once Daily as Oral Granules in Children Aged 3 to 6 Months
Brief Title: PK Study in 3- to 6- Month-Old Children (0476-268)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-268; 2006_545
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Montelukast sodium (Experimental): Participants receive montelukast sodium for 14 days.
  Interventions: Drug: MK-0476, montelukast sodium

INTERVENTIONS:
Drug: MK-0476, montelukast sodium — Duration of Treatment: 14 Days

SUMMARY:
The purpose of this study is to look at the preliminary safety profile of an investigational drug in children 3 to 6 months of age with bronchiolitis.

ELIGIBILITY:
Inclusion Criteria :

* Active bronchiolitis or a history of bronchiolitis and asthma-like symptoms

Exclusion Criteria :

* A history of any significant illness that will pose additional risk to the patient

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2003-07; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of montelukast oral granules in children aged 3 to 6 months. | 14 days

SECONDARY OUTCOMES:
To estimate the single-dose population pharmacokinetics, maximum plasma concentration, time to maximum plasma concentration, and apparent half-life of montelukast 4-mg oral granules in children aged 3 to 6 months. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Knorr B, Maganti L, Ramakrishnan R, Tozzi CA, Migoya E, Kearns G. Pharmacokinetics and safety of montelukast in children aged 3 to 6 months. J Clin Pharmacol. 2006 Jun;46(6):620-7. doi: 10.1177/0091270006288324. PMID 16707408